CLINICAL TRIAL: NCT07280273
Title: Effectiveness of Pain Science Education (PSE) in Patients With Fibromyalgia Syndrome (FMS) Living in Rural Areas.: a Randomized Clinical Trial.
Brief Title: Effectiveness of Pain Science Education in Patients With Fibromyalgia Syndrome Living in Rural Areas.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: María Catalina Osuna Pérez (Other)
Responsible Party: Sponsor-Investigator, María Catalina Osuna Pérez, Full professor at the university, University of Jaén
Organization: University of Jaén (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSE-RURAL
Record Dates: First submitted 2025-11-27; First posted 2025-12-12 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia Syndrome
Keywords: Fibromyalgia Syndrome; Pain Science Education
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSE group (Experimental)
  Interventions: Procedure: Pain Science Education
- Control group (No Intervention)

INTERVENTIONS:
Procedure: Pain Science Education — The intervention group will receive two 90-minute in-person Pain Education sessions, each delivered one week apart. The intervention will be delivered by a therapist experienced in educational interventions. The session content will be based on the most recent literature, clinical practice guidelines, and published literature on pain science, addressing concepts in a simple way so that patients can integrate them into their daily lives, with the goal of changing their knowledge and beliefs about pain. Images and metaphors will be used, avoiding the use of technical language to ensure knowledge transfer. After each session, any questions that may have arisen will be addressed. Participants will be given a dossier containing the session content to reinforce and integrate the knowledge acquired during the sessions, without providing additional information.
  Arms: PSE group

SUMMARY:
Fibromyalgia Syndrome (FMS) is a complex chronic pain disorder characterized by widespread pain associated with numerous symptoms. It is more common in women over 50 years of age with low educational and socioeconomic status living in rural areas. Pain Science Education (PSE) is one of the most widely used treatments for chronic pain management. This treatment consists of an educational intervention aimed at reconceptualizing and modifying erroneous cognitions regarding pain in these patients.

The objective of this study is to evaluate the effectiveness of PSE in patients with FMS living in rural areas. They will be randomly assigned to one of two treatment groups. The intervention group will receive two adapted in-person sessions (90 minutes per session/week) by a therapist experienced in teaching PSE. The control group will begin the conventional treatment they received before participating in the study. After the end of the study, patients in the control group will be given their intervention group records. The variables measured will include the impact of FMS on daily life, pain sensitivity, central sensitization, pain catastrophizing, fear of movement, anxiety and depression, self-efficacy, and assessment of knowledge and beliefs about PSE. Assessments will be conducted before the intervention, after the second PSE session, and three months later by the same researcher.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FM that meets the 2016 American College of Rheumatology (ACR) diagnostic criteria.
* Residence in a rural area of the province of Jaén (Spain).
* Age between 18 and 65 years.
* Spanish reading ability.
* Understanding and acceptance of the informed consent form to participate in the study.

Exclusion Criteria:

* -Patients diagnosed with any mental illness that prevents adherence to the intervention.
* Patients diagnosed with inflammatory rheumatic disease.
* Having a scheduled surgical intervention during the data collection process that could interfere with the results.
* Being pregnant or breastfeeding.
* Modification of pharmacological treatment during the study or in the last three months before the intervention.

These criteria have been established from a review of other clinical trials conducted with similar interventions in patients with FMS.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Pain sensitivity | All outcomes will be measured at the beginning of the study, at the end of all PSE sessions, and at the three-month follow-up.
  ain sensitivity was measured with the Pain Sensitiv-ity Questionnaire (PSQ), which consists of 17 items in a11-point Likert format. This questionnaire assesses painsensitivity based on pain intensity ratings (range: 0---10)of painful situations that occur in daily life. The PSQ canbe calculated as a total score (PSQ-total), a PSQ mod-erate score (the sum of items 1, 2, 4, 8, 15, 16 and17, which represent situations of moderate pain), or aPSQ minor score (the sum of items 3, 6, 7, 10, 11, 12and 14, which represent situations of mild pain). Items5, 9 and 13 are not taken into consideration becausethey represent non-painful situations. The Spanish vali-dation results showed an excellent internal consistency(Cronbach's ˛ > 0.9) and a substantial reliability (IntraclassCorrelation Coefficient > 0.8).
Impact of FMS on daily life | All outcomes will be measured at the beginning of the study, at the end of all PSE sessions, and at the three-month follow-up.
  To assess the impact of FMS on daily life, the Spanishversion of the revised Fibromyalgia Impact Questionnaire(FIQ) was used. It assesses the function, impact and symp-toms related to FMS and scores from 0 to 100, with100 being the maximum impact of FMS on QoL. TheSpanish FIQR had high internal consistency (Cronbach's ˛0.91---0.95). The test---retest reliability was good for theFIQR total score and its function and symptoms domains(intraclass correlation coefficient (ICC > 0.70), but modestfor the overall impact domain (ICC = 0.51).
Central sensitization | All outcomes will be measured at the beginning of the study, at the end of all PSE sessions, and at the three-month follow-up.
  Central sensitization (CS) was measured with the Span-ish version of the Central Sensitization Inventory (CSI).It is a self-report outcome measure designed to identifypatients who have symptoms that may be related to CSor CS syndromes such as FMS. It consists of 25 questionsrelated to common CS symptoms, with total scores rangingfrom 0 to 100. The Spanish version of the CSI demonstratedhigh internal consistency (Cronbach's ˛ = 0.872) and a one-dimensional factor structure.
Pain catastrophizing | All outcomes will be measured at the beginning of the study, at the end of all PSE sessions, and at the three-month follow-up.
  The Spanish version of the Pain Catastrophizing Scale (PCS) will be used to assess catastrophic thoughts about pain. This scale consists of 3 subscales graded from 0 (no negative thoughts or feelings) to 3 (maximum negative thoughts or feelings). It consists of 13 items with a 5-point Likert-type response scale (0 = Not at all; 4 = All the time), with a theoretical range of 0 to 52 points. Higher scores indicate a greater presence of catastrophic thoughts (43). It showed adequate internal consistency (Cronbach's α = 0.79), test-retest reliability (ICC = 0.84) and sensitivity to change (effect size ≥ 2). It is considered useful for clinical practice and research, having been carried out on a sample of 230 Spanish patients with FM.
Fear of Movement | All outcomes will be measured at the beginning of the study, at the end of all PSE sessions, and at the three-month follow-up.
  This will be assessed with the short version of the Tampa Kinesiophobia Scale (TSK-11). This is one of the most widely used measures for assessing pain-related fear in patients with pain. It is an 11-item self-report measure of fear of movement and re-injury, rated on a four-point scale from "strongly agree" to "strongly disagree." The total score ranges from 11 to 44. Ratings are summed to obtain a total score, with higher scores indicating greater fear of re-injury. This Spanish version demonstrated good internal consistency (Cronbach's α = 0.79) and moderate test-retest reliability (r = 0.55).
Anxiety and depression | All outcomes will be measured at the beginning of the study, at the end of all PSE sessions, and at the three-month follow-up.
  Anxiety and depression were assessed using the Span-ish version of the Hospital Anxiety and Depression Scale(HADS). This scale comprises two subscales: the HAD Anx-iety subscale (HADA) and the HAD Depression subscale(HADD). This questionnaire consists of 14 items, ratedfrom 0 (no distress) to 3 (maximum distress). The cut-offscore for the presence of anxiety and depression symp-toms must be equal to or greater than 8. The internalconsistency of the scales of the Spanish version is Cron-bach's ˛ = 0.80 for the HADA and Cronbach's ˛ = 0.85 forthe HADD.
Self-efficacy | All outcomes will be measured at the beginning of the study, at the end of all PSE sessions, and at the three-month follow-up.
  This will be assessed using the Spanish adaptation of the Chronic Pain Self-Efficacy Scale. The total score, obtained from the summation of the responses to the 19 items comprising the questionnaire, will be used. The subject must answer the degree to which they consider themselves capable of performing certain activities or managing their pain, emotional problems, or other symptoms associated with chronic pain. Responses are made using a Likert-type scale from 0 (I feel totally incapable) to 10 (I see myself as totally capable), with a theoretical range of 0 to 190. High scores indicate a high perception of self-efficacy. It is considered an appropriate instrument for assessing self-efficacy expectations in patients with chronic pain of benign origin. This scale presented good psychometric properties in terms of reliability and construct validity, presenting a high internal consistency (Cronbach's α = 0.91) and a high test-retest reliability (ICC = 0.75) for the total
Knowledge and beliefs about PSE | All outcomes will be measured at the beginning of the study, at the end of all PSE sessions, and at the three-month follow-up.
  Knowledge and beliefs about PSE: This will be assessed using the Pain Concept Questionnaire (COPI-Adult). It is unidimensional and consists of 13 items. It has acceptable internal consistency (α=0.78) and good test-retest reliability at one week (Intraclass Correlation Coefficient=0.84 (95% confidence interval: 0.71-0.91).

CONTACTS AND LOCATIONS:
Overall Officials: María Catalina Osuna-Pérez, PhD, Principal Investigator — University of Jaén; Noelia Zagalaz Anula, PhD, Principal Investigator — University of Jaén
Locations (1):
- Fisio Mas, Peal de Becerro, Jaén, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salazar-Mendez J, Nunez-Cortes R, Suso-Marti L, Ribeiro IL, Garrido-Castillo M, Gacitua J, Mendez-Rebolledo G, Cruz-Montecinos C, Lopez-Bueno R, Calatayud J. Dosage matters: Uncovering the optimal duration of pain neuroscience education to improve psychosocial variables in chronic musculoskeletal pain. A systematic review and meta-analysis with moderator analysis. Neurosci Biobehav Rev. 2023 Oct;153:105328. doi: 10.1016/j.neubiorev.2023.105328. Epub 2023 Jul 27. PMID 37516218
- [Background] Ceballos-Laita L, Mingo-Gomez MT, Navas-Camara F, Estebanez-de-Miguel E, Caudevilla-Polo S, Verde-Rello Z, Fernandez-Araque A, Jimenez-Del-Barrio S. Therapeutic Exercise and Pain Neurophysiology Education in Female Patients with Fibromyalgia Syndrome: A Feasibility Study. J Clin Med. 2020 Nov 5;9(11):3564. doi: 10.3390/jcm9113564. PMID 33167469
- [Background] Boomershine CS. Fibromyalgia: the prototypical central sensitivity syndrome. Curr Rheumatol Rev. 2015;11(2):131-45. doi: 10.2174/1573397111666150619095007. PMID 26088213
- [Background] Sauch Valmana G, Miro Catalina Q, Carrasco-Querol N, Vidal-Alaball J. Gender, Mental Health and Socioeconomic Differences in Fibromyalgia: A Retrospective Cohort Study Using Real-World Data from Catalonia. Healthcare (Basel). 2023 Feb 10;11(4):530. doi: 10.3390/healthcare11040530. PMID 36833067
- [Background] Catala P, Blanco S, Perez-Calvo S, Luque-Reca O, Bedmar D, Penacoba C. Does the Rural Environment Influence Symptomatology and Optimize the Effectiveness of Disease Acceptance? A Study Among Women With Fibromyalgia. Front Psychol. 2021 Apr 29;12:658974. doi: 10.3389/fpsyg.2021.658974. eCollection 2021. PMID 33995219
- [Background] Font Gaya T, Bordoy Ferrer C, Juan Mas A, Seoane-Mato D, Alvarez Reyes F, Delgado Sanchez M, Martinez Dubois C, Sanchez-Fernandez SA, Marena Rojas Vargas L, Garcia Morales PV, Olive A, Rubio Munoz P, Larrosa M, Navarro Ricos N, Sanchez-Piedra C, Diaz-Gonzalez F, Bustabad-Reyes S; Working Group Proyecto EPISER2016. Prevalence of fibromyalgia and associated factors in Spain. Clin Exp Rheumatol. 2020 Jan-Feb;38 Suppl 123(1):47-52. Epub 2020 Jan 8. PMID 31928589
- [Background] Bidonde J, Busch AJ, Schachter CL, Webber SC, Musselman KE, Overend TJ, Goes SM, Dal Bello-Haas V, Boden C. Mixed exercise training for adults with fibromyalgia. Cochrane Database Syst Rev. 2019 May 24;5(5):CD013340. doi: 10.1002/14651858.CD013340. PMID 31124142
- [Background] Al Sharie S, Varga SJ, Al-Husinat L, Sarzi-Puttini P, Araydah M, Bal'awi BR, Varrassi G. Unraveling the Complex Web of Fibromyalgia: A Narrative Review. Medicina (Kaunas). 2024 Feb 4;60(2):272. doi: 10.3390/medicina60020272. PMID 38399559
- [Background] Queiroz LP. Worldwide epidemiology of fibromyalgia. Curr Pain Headache Rep. 2013 Aug;17(8):356. doi: 10.1007/s11916-013-0356-5. PMID 23801009